CLINICAL TRIAL: NCT00452296
Title: Tight Glycemic Control in Acute Exacerbations of COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Idit F Liberty, Dr Idit Liberty MD, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: sor450807ctil
Record Dates: First submitted 2007-03-25; First posted 2007-03-27 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: COPD; Hyperglycemia
Keywords: inpatients with COPD; glucose control
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tight insulin treatment in patients hospitalized with COPD exacerbation — treatment with basal plus bolus insulin
Procedure: tight glycemic control — treatment with basal and bolus insulin

SUMMARY:
Glucose control has been shown as an important and independent prognostic factor in several acute conditions in hospitalized patients, including Acute MI, stroke, cardiac surgery and in critical care units.

Patients with acute exacerbation of COPD (AECOPD)and diabetes treated with insulin had a longer in-patient stay and more frequent isolation of Gram negative bacteria from sputum than those without diabetes.Hyperglycemia (>11 mmol/l) on admission predicted failure of non-invasive ventilation and infectious pulmonary complications in patients admitted to the ICU with acute respiratory failure caused by severe AECOPD.

The primary goal of this study is to test the hypothesis that in AECOPD, tight glycemic control during hospital stay will improve outcome of hospitalization.

The secondary goal of this study is to test new ways in controlling patients in the internal medicine ward.

ELIGIBILITY:
Inclusion Criteria:

* current or past smokers (at least 20 py)
* patient with COPD be ATS criteria
* hospitalized with acute exacerbation, 2/3 criteria:1- worsening of SOB 2-change in sputum volume 3- change in sputum color
* signed informed concent

Exclusion Criteria:

* respiratory failure (pH<7.35 ו Pco2>60 )
* pneumonia
* pneumothorax
* bronchiectasis
* lung collapse
* congestive heart failure
* lung cancer
* suspected pulmonary emboli
* immune deficiency (acquired 0r congenital)
* cystic fibrosis
* post lung implantation
* asthma/ non smokers

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
mortality | one year

SECONDARY OUTCOMES:
hospialization | one year

CONTACTS AND LOCATIONS:
Overall Officials: Idit F Liberty, Principal Investigator — Soroka University Medical Center